CLINICAL TRIAL: NCT02204761
Title: Definitive Re-irradiation With Proton Beam Radiotherapy for Patients With Recurrent Thoracic Cancers
Brief Title: Proton Beam Re-Irradiation in Thoracic Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Zeng, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9148; NCI-2014-01468 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9148 (Other: University of Washington); P30CA015704 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Malignant Neoplasm in the Lung; Recurrent Disease; Thoracic Neoplasm
MeSH Terms: conditions — Recurrence; Thoracic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Proton beam radiation therapy
  Interventions: Radiation: Proton Beam Radiation Therapy

INTERVENTIONS:
Radiation: Proton Beam Radiation Therapy — Undergo proton beam re-irradiation therapy

SUMMARY:
This pilot clinical trial studies proton beam radiation therapy in treating patients with thoracic cancer that has come back and have received prior radiation therapy. Proton beam radiation therapy uses high energy protons to kill tumor cells and may cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the grade 3 toxicity associated with thoracic re-irradiation with proton therapy, with prospectively applied normal organ radiation dose limits.

SECONDARY OBJECTIVES:

I. To assess the efficacy of thoracic re-irradiation with proton therapy.

OUTLINE:

Patients undergo proton beam radiation therapy per standard of care.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Women of child-bearing age must have a negative pregnancy test
* Patients must have received prior radiation treatment to the chest; records of prior radiation treatment must be available
* Patients must have received prior chest radiation at least 3 months prior to enrollment in this trial; radiation treatment to other body sites not overlapping with current radiation fields are allowed within the 3 months period (example, brain radiation is allowed)
* Patients must have a prior diagnosis of cancer inside the thoracic cavity; both primary thoracic malignancies (such as lung cancer) as well as metastatic lesions (such as metastatic breast cancer or colorectal cancer to the lungs) are allowed; patient must have pathologic confirmation of the recurrent thoracic tumor, or have an enlarging thoracic mass (as seen on two computed tomography [CT] scans at least 6 weeks apart, with either a > 25% or > 5 mm increase in longest dimension)
* Patients must have a life expectancy of > 6 months
* Patients must have measurable disease to be treated with proton radiation (minimum tumor dimension at least 10 mm on CT imaging)
* Patients should have either non-metastatic cancer of the thorax, or metastatic cancer to the thorax and candidate for definitive radiation dose to the thoracic tumor (not palliative intent), tumor radiation dose to at least BED2Gy 60 Gy
* Patients must be able to receive proton radiation treatment
* All stages of cancer are eligible
* There are no limits on prior therapy; patients are allowed to have prior chemotherapy and surgery; patients are allowed to have concurrent chemotherapy with radiation treatment; patients are allowed to have chemotherapy or surgery after radiation treatment
* Patients are allowed to be on another study concurrent with this protocol
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have never received radiation to the chest
* Patients who received radiation to the chest within the past 3 months (in a region that overlaps with current radiation fields)
* Patients with life expectancy < 6 months
* Pregnant women
* Patients unable to provide informed consent
* Prisoners

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - ProCure Proton Therapy Center-Seattle, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Proton Beam Radiation Therapy): Patients undergo proton beam radiation therapy per standard of care.
  Proton Beam Radiation Therapy: Undergo proton beam radiation therapy
Period: Overall Study
Arm/Group | Treatment (Proton Beam Radiation Therapy)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Proton Beam Radiation Therapy)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Number of participants with Grade 3+ toxicity from radiation [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Greater Toxicity Attributable to Radiation Treatment
Description: Toxicity will be graded based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 3 generally means hospitalization required for management of side effects.
Time Frame: Up to 3 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Proton Beam Radiation Therapy)
Number analyzed (Participants) | 6
Participants | 2

2. Secondary Outcome: Number of Participants With Grade 2 Toxicity Attributable to Radiation Treatment
Description: Toxicity will be graded based on Common Terminology Criteria for Adverse Events (CTCAE) v 4.0. Grade 2 generally means medical therapy required to intervene due to toxicity.
Time Frame: Up to 3 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Proton Beam Radiation Therapy)
Number analyzed (Participants) | 6
Participants | 2

3. Secondary Outcome: Number of Participants With Local Control of Cancer
Description: Number of participants who did not have local failure as defined by: tumor progression per Response Evaluation Criteria in Solid Tumors criteria - at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions inside the full dose radiation field.
Time Frame: Up to 3 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Proton Beam Radiation Therapy)
Number analyzed (Participants) | 6
Participants | 6

4. Secondary Outcome: Number of Participants Alive
Description: Number of participants alive.
Time Frame: Up to 3 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Proton Beam Radiation Therapy)
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment (Proton Beam Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Proton Beam Radiation Therapy) (N=6)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02204761/Prot_SAP_000.pdf